CLINICAL TRIAL: NCT02535507
Title: Single Arm Phase II Clinical Trial to Investigate the Efficacy and Safety of Pyrotinib as a Single Agent in HER2 Mutation Advanced Non-small Cell Lung Cancer Patients Who Failed to Previous at Least 2nd Line Treatments
Brief Title: Efficacy and Safety of Pyrotinib in Patients With HER2 Mutation Advanced Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Caicun Zhou, MD,PhD, Tongji University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FK1406
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: pyrotinib; HER2; Non-small Cell Lung Cancer; Phase II
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pyrotinib treatment arm (Experimental): pyrotinib treatment arm
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — Drug: Pyrotinib pyrotinib, single agent, 400mg p.o once daily until disease progressed

SUMMARY:
Various driver gene mutations have been identified in lung cancer. Among them, human epidermal growth factor 2 (HER2) was identified in about approximately 2% of non-small cell lung cancers.Pyrotinib is an oral tyrosine kinase inhibitor targeting both HER-1 and HER-2 receptors. This study is designed to evaluate the efficacy and safety of Pyrotinib in patients with HER2 positive advanced Non-small cell lung cancer.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy and safety of Pyrotinib in patients with HER2 positive advanced pre-treated Non-small cell lung cancer.

To observe objective response rate (ORR) of pyrotinib in HER2 positive NSCLC. To observe Progression free survival （PFS）. To assess the overall survival (OS). To assess side effects. To evaluate quality of life. To explore the relationship between biomarkers and the toxicity/efficacy of Pyrotinib.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 and ≤80 years.
* ECOG performance status of 0 to 1.
* Life expectancy of more than 12 weeks.
* At least one measurable lesion exists.(RECIST 1.1)
* Histologically or cytologic confirmed HER2 positive advanced Non-small cell lung cancer who failed prior therapies.
* Required laboratory values including following parameters:

ANC: ≥ 1.5 x 10^9/L, Platelet count: ≥ 80 x 10^9/L, Hemoglobin: ≥ 90 g/L, Total bilirubin: ≤ 1.5 x upper limit of normal, ULN, ALT and AST: ≤ 1.5 x ULN, BUN and creatine clearance rate: ≥ 50 mL/min LVEF: ≥ 50% QTcF: < 470 ms

* Signed informed consent.

Exclusion Criteria:

* Subjects with third space fluid that can not be controled by drainage or other methods.
* Subjects that are unable to swallow tablets, or dysfunction of gastrointestinal absorption.
* Less than 4 weeks from the last radiotherapy,chemotherapy,target therapy
* Subjects with uncontrolled hypokalemia and hypomagnesemia before study entry.
* Subjects who can not interrupt the using of the drugs that may cause QT prolongation during study.
* Receiving any other antitumor therapy.
* Known history of hypersensitivity to pyrotinib or any of it components. Ongoing infection (determined by investigator).
* History of immunodeficiency, including HIV-positive, suffering from other acquired, congenital immunodeficiency disease, or history of organ transplantation.
* Subjects had any heart disease, including: (1) angina; (2) requiring medication or clinically significant arrhythmia; (3) myocardial infarction; (4) heart failure; (5) Any heart diseases judged by investigator as unsuitable to participate in the trial.
* Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test.
* Known history of neurological or psychiatric disease, including epilepsy or dementia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | tumor assessment every 6-8 weeks after the initiation of pyrotinib, up to 24 months
  To evaluate objective response rate 6-8 weeks after the initiation of pyrotinib

SECONDARY OUTCOMES:
Progression Free Survival | 24 months
  PFS is evaluated in 24 months since the treatment began

OTHER OUTCOMES:
overall survival | 24 months
  evaluated in the 24th month since the treatment began
Safety and Tolerability | 24 months
  Number of Participants with treatment related Adverse Events as Assessed by CTCAE v4.0
quality of life (measured by questionnaire) | 24 months
  Change from baseline in Pain on the 11 point short pain scale (SPS-11)

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD,PhD, Principal Investigator — Shanghai Pulmonary Hospital, Tongji University
Locations (1):
- Department of Oncology, Shanghai pulmonary hospital, Shanghai, China

REFERENCES:
- [Derived] Mao S, Yang S, Liu X, Li X, Wang Q, Zhang Y, Chen J, Wang Y, Gao G, Wu F, Jiang T, Zhang J, Yang Y, Lin X, Zhu X, Zhou C, Ren S. Molecular correlation of response to pyrotinib in advanced NSCLC with HER2 mutation: biomarker analysis from two phase II trials. Exp Hematol Oncol. 2023 Jun 9;12(1):53. doi: 10.1186/s40164-023-00417-y. PMID 37296463
- [Derived] Wang Y, Jiang T, Qin Z, Jiang J, Wang Q, Yang S, Rivard C, Gao G, Ng TL, Tu MM, Yu H, Ji H, Zhou C, Ren S, Zhang J, Bunn P, Doebele RC, Camidge DR, Hirsch FR. HER2 exon 20 insertions in non-small-cell lung cancer are sensitive to the irreversible pan-HER receptor tyrosine kinase inhibitor pyrotinib. Ann Oncol. 2019 Mar 1;30(3):447-455. doi: 10.1093/annonc/mdy542. PMID 30596880